CLINICAL TRIAL: NCT03969992
Title: A Partially Blinded, Randomized, Controlled, Parallel-Group, Dose-Ranging Study to Determine the Efficacy, Safety and Tolerability of AeroFact in Preterm Infants at Risk of Worsening Respiratory Distress Syndrome
Brief Title: A Dose-Ranging Study to Determine the Efficacy, Safety and Tolerability of AeroFact
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerogen Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-AF-CLN-002
Record Dates: First submitted 2019-04-05; First posted 2019-05-31 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: Respiratory Distress Syndrome; BPD; surfactant; Preterm Infant
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — SF-RI 1, bovine surfactant preparation

STUDY DESIGN:
Intervention Model Description: Partially Blinded, Randomized, Parallel-Group Dose Ranging
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking within active arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- nCPAP alone (Other): Standard of Care (nasal continuous positive airway pressure-nCPAP) with instilled bolus surfactant when medically necessary
  Interventions: Other: nCPAP
- Drug: Low Dose AeroFact (Experimental): AeroFact-low dose SF-RI 1
  Interventions: Drug: AeroFact
- Drug: High Dose AeroFact (Experimental): AeroFact-high dose SF-RI 1
  Interventions: Drug: AeroFact

INTERVENTIONS:
Drug: AeroFact — Aerosolized SF-RI 1
  Other Names: SF-RI 1
  Arms: Drug: High Dose AeroFact; Drug: Low Dose AeroFact
Other: nCPAP — nCPAP (nasal continuous positive airway pressure) alone
  Arms: nCPAP alone

SUMMARY:
The purpose of this two-part Phase 2 study is to assess the safety, tolerability and efficacy of aerosolized SF-RI 1 (AeroFact) when delivered via nCPAP at two different doses.

DETAILED DESCRIPTION:
Part I Primary Objective To determine an optimal dose of AeroFact administered by nasal continuous positive airway pressure (nCPAP) versus stand of care in reducing the rate of intubation/cannulation and bolus surfactant instillation in the first 7 days after birth.

Part II Primary Objective To evaluate pulmonary outcomes and respiratory utilization at 3, 6, 9, and 12 months post-menstrual age (PMA)

ELIGIBILITY:
Inclusion Criteria:

1. Parental consent obtained prior to study procedures being performed (pre-natal consent is allowed)
2. 26 0/7 to 30 6/7 weeks of gestational age
3. Weight <2.0 Kg
4. Respiratory Severity Score (RSS) 1.4-2.0

Exclusion Criteria:

1. Apgar score less than or equal to 5 at five minutes after birth
2. Need for chest compressions or administration of epinephrine or bicarbonate in the delivery room
3. Premature rupture of membranes (PROM) > 14 days
4. Need for intubation and/or mechanical ventilation prior to enrollment
5. Active pneumothorax requiring chest tube
6. Significant congenital anomaly, chromosomal abnormality
7. Concomitant treatments with inhaled nitric oxide

Ages: 26 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Durand, MD, Study Director — Aerogen Pharma Corp
Locations (41):
- United States (37):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit, Berkeley, California
  - Children's Hospital Orange County, Orange, California
  - University of Colorado, Aurora, Colorado
  - University of Florida Health, Jacksonville, Florida
  - Wolfson Children's Hospital, Jacksonville, Florida
  - South Miami Hospital, Miami, Florida
  - Advent Health, Orlando, Florida
  - Winnie Palmer Hospital, Orlando, Florida
  - Northside Hospital Atlanta, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Hospital of South Bend, South Bend, Indiana
  - University of Louisville, Louisville, Kentucky
  - Barbara Bush Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Children's and Women's (C & W) Mott Hospital, Ann Arbor, Michigan
  - Children's Health Care d/b/a Children's Minnesota, Minneapolis, Minnesota
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Maimonides Hospital, Brooklyn, New York
  - Mount Sinai Kravis Children's Hospital, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - NY Presbyterian Morgan Stanley Children's Hospital-Columbia, New York, New York
  - West Chester Medical Center-Maria Fareri Children's Hospital, Valhalla, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Grant Hospital, Columbus, Ohio
  - Texas Health-Methodist Harris, Fort Worth, Texas
  - Women's Hospital of Texas, Houston, Texas
  - Children's Hospital of San Antonio (CHofSA), San Antonio, Texas
  - Methodist Children's Hospital, San Antonio, Texas
  - North Central Baptist Hospital, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- Canada (4):
  - IWK Hospital, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Mt. Sinai Hospital, Toronto, Ontario
  - CHU de Québec-Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: nCPAP Alone: nCPAP (nasal continuous positive airway pressure) alone
- Drug: Low Dose AeroFact: AeroFact 108 mg/kg/dose
- Drug: High Dose AeroFact: AeroFact 216 mg/kg/dose
Period: Part 1: Birth to Discharge/40 Weeks PMA
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Started | 92 | 83 | 86
Completed | 89 | 80 | 81
Not Completed | 3 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Death | 2 | 3 | 2
Period: Part 2: Discharge/40 Wks PMA to 12 Mos
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Started | 89 | 80 | 81
Completed | 74 | 71 | 71
Not Completed | 15 | 9 | 10
Not completed — Lost to Follow-up | 12 | 8 | 9
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients were included in the ITT and Safety analysis populations, regardless of whether or not they received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact | Total
Number analyzed (Participants) | 92 | 83 | 86 | 261
Age, Continuous [Mean (Standard Deviation); unit: weeks gestational age] — Gestational age in weeks
  weeks gestational age | 29.2 (1.3) | 29.1 (1.4) | 29.1 (1.5) | 29.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 38 | 37 | 122
  Male | 45 | 45 | 49 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 22 | 12 | 47
  Not Hispanic or Latino | 77 | 58 | 72 | 207
  Unknown or Not Reported | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 1 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 12 | 15 | 43
  White | 57 | 50 | 48 | 155
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 16 | 20 | 14 | 50
Birth weight [Mean (Standard Deviation); unit: grams] | 1195.1 (297.9) | 1245.1 (301.5) | 1248.7 (303.9) | 1228.7 (300.9)
Vaginal delivery [Count of Participants; unit: Participants] | 14 | 25 | 19 | 58
Multiple gestation [Count of Participants; unit: Participants] | 30 | 29 | 26 | 85
Age at Randomization [Mean (Standard Deviation); unit: hours] | 10.0 (7.2) | 8.2 (6.5) | 8.9 (6.9) | 9.1 (6.9)
FiO2 at Randomization [Mean (Standard Deviation); unit: Percentage of inspired oxygen] — Fraction of inspired oxygen; Higher scores indicate more supplemental oxygen was needed
  Percentage of inspired oxygen | 0.27 (0.05) | 0.27 (0.04) | 0.27 (0.05) | 0.27 (0.05)
Respiratory Severity Score at Randomization [Mean (Standard Deviation); unit: units on a scale] — mean airway pressure [MAP] × FiO2; Higher scores suggest greater breathing difficulty
  units on a scale | 1.7 (0.2) | 1.7 (0.2) | 1.7 (0.3) | 1.7 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Intubation/Cannulation and Instilled Surfactant
Description: Number of patients who require intubation/cannulation with bolus surfactant instillation
Time Frame: First 7 days of life
Population: Per Protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Number analyzed (Participants) | 89 | 68 | 70
Participants | 45 | 21 | 26
Statistical Analysis 1: Comparison: Control: nCPAP Alone vs Drug: Low Dose AeroFact vs Drug: High Dose AeroFact; Test type: Superiority; p = 0.1924, Generalized estimating equation method — A closed test procedure is used to protect the type I error rate; the order of testing was: AeroFact high dose compared to control and if significant (p-value <0.05), the AeroFact low dose was compared to the control

2. Secondary Outcome: Time to First Intubation/Cannulation and Bolus Surfactant Instillation
Description: Time from randomization to intubation/cannulation and bolus surfactant instillation in the first 7 days of life
Time Frame: First 7 days of life
Population: Per protocol population
Measure: Median (Full Range); unit: hours
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Number analyzed (Participants) | 45 | 21 | 26
hours | 17.5 [2.0 to 53.9] | 13.6 [3.2 to 43.4] | 22.4 [1.8 to 53.7]

3. Secondary Outcome: Proportion of Infants Who Received Multiple Doses of Bolus Surfactant
Time Frame: First 7 days of life
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Number analyzed (Participants) | 89 | 68 | 70
Participants | 7 | 1 | 5

4. Secondary Outcome: Number of Days on Invasive Mechanical Ventilation
Description: Total number of days each participant required support with invasive mechanical ventilation
Time Frame: Assessed daily from birth to 40 weeks post-menstrual age or discharge
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Number analyzed (Participants) | 44 | 28 | 28
Days | 4.8 (7.1) | 6.0 (16.7) | 4.0 (4.7)

5. Secondary Outcome: Proportion of Patients Survived Without Bronchopulmonary Dysplasia (BPD) at 36 Weeks Post-menstrual Age (PMA)
Description: Total number of patients per treatment group who were alive and did not experience BPD at 36 weeks PMA
Time Frame: Birth to 36 weeks post-menstrual age
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Number analyzed (Participants) | 89 | 68 | 70
Participants | 69 | 55 | 53

6. Secondary Outcome: Proportion of Patients Survived Without Bronchopulmonary Dysplasia (BPD) at 40 Weeks Post-menstrual Age (PMA)
Description: Total number of patients per treatment group who were alive and did not experience BPD at 40 weeks PMA
Time Frame: Birth to 40 weeks post-menstrual age
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
Number analyzed (Participants) | 89 | 68 | 70
Participants | 74 | 58 | 56

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from randomization through NICU discharge or 40 weeks post-menstrual age (PMA) in Part 1. Only fatal SAEs were collected for up to 12 months in Part 2.
Arm/Group | Control: nCPAP Alone | Drug: Low Dose AeroFact | Drug: High Dose AeroFact
All-Cause Mortality (participants affected / at risk) | 2/92 | 3/83 | 2/86
Serious Adverse Events (participants affected / at risk) | 7/92 | 9/83 | 5/86
Other Adverse Events (participants affected / at risk) | 43/92 | 45/83 | 42/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control: nCPAP Alone (N=92) | Drug: Low Dose AeroFact (N=83) | Drug: High Dose AeroFact (N=86)
Necrotizing enterocolitis neonatal (Gastrointestinal disorders) | 2 | 2 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 2 | 0
Meconium ileus (Gastrointestinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Pulmonary hemorrhage neonatal (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Intraventricular hemorrhage neonatal (Nervous system disorders) | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control: nCPAP Alone (N=92) | Drug: Low Dose AeroFact (N=83) | Drug: High Dose AeroFact (N=86)
Intraventricular hemorrhage neonatal (Nervous system disorders) | 6 | 15 | 18
Retinopathy or prematurity (Eye disorders) | 14 | 13 | 13
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4
Infantile apnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary hemorrhage neonatal (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 11 | 5 | 4
Necrotizing enterocolitis neonatal (Gastrointestinal disorders) | 5 | 5 | 5
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 3 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1 | 1
Sepsis (Infections and infestations) | 4 | 5 | 3
Bradycardia neonatal (Cardiac disorders) | 2 | 6 | 1
Patent ductus arteriosus repair (Surgical and medical procedures) | 4 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03969992/Prot_SAP_000.pdf